CLINICAL TRIAL: NCT04533880
Title: The Effect of Bone-void Filler on Anterior Knee Pain Following ACL Reconstruction With Bone-Patellar Tendon Bone Autograft
Brief Title: The Effect of Bone-void Filler on Anterior Knee Pain Following ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00081
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: ACL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control (Placebo Comparator): The control group will receive autologous bone obtained from the BTBPB graft harvest
  Interventions: Other: Autologous bone graft
- Autologous Bone + DBM (Active Comparator): Autologous bone plus demineralized bone matrix
  Interventions: Device: DBM; Other: Autologous bone graft
- Autologous Bone + Calcium Phosphate Cement (Active Comparator): Autologous bone plus calcium phosphate cement
  Interventions: Device: Calcium phosphate cement; Other: Autologous bone graft

INTERVENTIONS:
Device: DBM — Demineralized bone matrix (Allosync, CDMB Putty, Arthrex, Naples, FL)
  Arms: Autologous Bone + DBM
Device: Calcium phosphate cement — Quickset, Arthrex, Naples, FL
  Arms: Autologous Bone + Calcium Phosphate Cement
Other: Autologous bone graft — Autologous bone grafting involves utilizing bone obtained from the same individual receiving the graft

SUMMARY:
One of the common complaints after ACLR with BPTB autograft anterior knee pain. It is thought that this may be due to harvesting the patellar tendon for graft use. Specifically, this may be due to the bone defect that is left after graft harvesting. There is currently no consensus on a gold standard for treating the bone defect with surgeons using multiple commercially available bone void fillers as well as autologous bone graft in standard practice.

The purpose of the proposed study is to evaluate the effect bone-void filler on anterior knee pain following ACL reconstruction BPTB autograft.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACLR with BPTB autograft
* Skeletally mature (as defined by closed growth plates on plain radiograph)
* At least 18 years of age
* Willing and able to provide consent

Exclusion Criteria:

* knee with intact ACL
* skeletally immature (as defined by open physis on plain radiograph)
* pregnant
* less than 18 years of age
* previous ACL repair or reconstruction
* unable to speak english or perform informed consent
* multiligamentous knee injury (two or more ligaments requiring surgical attention)
* varus or valgus malalignment greater than 3 degrees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strauss, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Orthopedic Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be provided upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to eric.strauss@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement
Started | 52 | 50 | 48
Completed | 52 | 49 | 47
Not Completed | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement | Total
Number analyzed (Participants) | 52 | 49 | 47 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (6.8) | 28.8 (8.1) | 28.8 (6.5) | 28.43 (7.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 27 | 71
  Male | 34 | 23 | 20 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 52 | 49 | 47 | 148
Region of Enrollment [Number; unit: participants]
  United States | 52 | 49 | 47 | 148

OUTCOME MEASURES:

1. Primary Outcome: Score on Knee Injury and Osteoarthritis Outcome Score (KOOS) Survey
Description: The KOOS survery comprises 42 questions; questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), quality of life (4 questions). Each item is rated on a Likert scale from 0 to 4. The score is calculated by summing the responses. The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain / higher difficulty in function.
Time Frame: Month 12 Post-Op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement
Number analyzed (Participants) | 52 | 49 | 47
score on a scale | 67 (6.1) | 69 (6.3) | 67.7 (8.2)

2. Primary Outcome: Score on Kujala Anterior Knee Pain Scale (AKPS)
Description: The Kujala AKPS is a 13-item screening instrument designed to assess patellofemoral pain in adolescents and young adults, with a variable ordinal response format. The total score is the sum of responses; total scores range from 0 to 100. Lower scores indicate greater signs of knee pain.
Time Frame: Month 12 Post-Op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement
Number analyzed (Participants) | 52 | 49 | 47
score on a scale | 87.1 (11) | 85.7 (17) | 86.2 (12.1)

3. Primary Outcome: Change in VAS Score for Anterior Knee Pain
Description: The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." The total score range is 0-100; the higher the score, the worse the pain.
Time Frame: Baseline, Month 12 Post-Op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement
Number analyzed (Participants) | 52 | 49 | 47
score on a scale | -5.5 (24.3) | -8.4 (26.9) | 1 (26.4)

ADVERSE EVENTS:
Time Frame: 12 months post-operation.
Description: Adverse event information collected at each study visit.
Arm/Group | Control | Autologous Bone + DBM | Autologous Bone + Calcium Phosphate Cement
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT04533880/Prot_SAP_000.pdf